CLINICAL TRIAL: NCT01181804
Title: A Definitive Bioequivalence Study of a New Boceprevir (SCH 503034) Tablet Formulation Compared to the Current Capsule Form in Healthy Male and Female Subjects.
Brief Title: Comparison of Safety and Resulting Blood Level Profiles After Administration of a New Boceprevir Tablet Versus Its Current Capsule Formulation for Treatment of Chronic Hepatitis C (P06992)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P06992
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
Keywords: boceprevir; hepatitis C; bioequivalence; SCH 503034
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Boceprevir Tablets then Capsules (fed) (Experimental): Participants will start therapy with a single dose of boceprevir tablets, orally, in fed condition, and then 4 days later will take a single dose of boceprevir capsules, orally, in fed condition.
  Interventions: Drug: boceprevir
- Boceprevir Capsules then tablets (fed) (Experimental): Participants will start therapy with a single dose of boceprevir capsules, orally, in fed condition, and then 4 days later will take a single dose of boceprevir tablets, orally, in fed condition.
  Interventions: Drug: boceprevir
- Boceprevir Tablets then Capsules (fasted) (Experimental): Participants will start therapy with a single dose of boceprevir tablets, orally, following an overnight fast, and then 4 days later will take a single dose of boceprevir capsules, orally, following an overnight fast.
  Interventions: Drug: boceprevir
- Boceprevir Capsules then Tablets (fasted) (Experimental): Participants on this study arm will start therapy with a single dose of boceprevir capsules, orally, following an overnight fast, and then 4 days later will take a single dose of boceprevir tablets, orally, following an overnight fast.
  Interventions: Drug: boceprevir

INTERVENTIONS:
Drug: boceprevir — Boceprevir (tablet or capsule) at 800 mg administered under either fed or fasted conditions.
  Other Names: SCH 503034
  Arms: Boceprevir Tablets then Capsules (fed)
Drug: boceprevir — Boceprevir (tablet or capsule) at 800 mg administered under either fed or fasted conditions.
  Other Names: SCH 503034
  Arms: Boceprevir Capsules then tablets (fed)
Drug: boceprevir — Boceprevir (tablet or capsule) at 800 mg administered under either fed or fasted conditions.
  Other Names: SCH 503034
  Arms: Boceprevir Tablets then Capsules (fasted)
Drug: boceprevir — Boceprevir (tablet or capsule) at 800 mg administered under either fed or fasted conditions.
  Other Names: SCH 503034
  Arms: Boceprevir Capsules then Tablets (fasted)

SUMMARY:
This is a single-dose, randomized, cross-sectional comparison study examining the relative safety and resulting blood level profiles after administration of a new boceprevir tablet formulation versus its current capsule formulation for treatment of chronic hepatitis C. In Part 1 of the study participants will receive boceprevir tablets and capsules under fed conditions. In Part 2 of the study a new group of participants will receive boceprevir tablets and capsules under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to give written informed consent for the trial and able to adhere to dose and visit schedules.
* Subjects must be willing to give written informed consent for pharmacogenetic

testing, and able to adhere to applicable visit schedules.

- Subjects of either gender and of any race between the ages of 18 and 65

years, inclusive, having a Body Mass Index (BMI) between 18 and 32,

inclusive. BMI = weight (kg)/height (m)^2. (Individuals with values outside (or

indicate lower or higher) of these ranges may be enrolled if clinically

acceptable to the investigator and sponsor.)

* Subjects' clinical laboratory tests (complete blood count [CBC], blood chemistry, and urinalysis) must be within normal limits or clinically acceptable to the investigator and within an allowed expanded range supplied by sponsor. However, subject's liver function test results (ie, aspartate aminotransferase [AST], alanine aminotransferase [ALT]) must not be elevated above normal limits at Screening and on Day -1. No rescreening of liver function tests will be allowed.
* Subjects must be free of any clinically significant disease that would interfere with the study evaluations.
* The Screening 12 lead electrocardiogram [ECG] conduction intervals must be within gender specific normal range (e.g, ECG QTcB,measure in males ≤430 msec and QTcB measure in females ≤450 msec, PR interval ≤200 msec).
* Vital sign measurements (taken after ~3 minutes in a sitting position) must be

within the following ranges: (Individuals with values outside of these ranges

may be enrolled if clinically acceptable to the investigator and sponsor.)

1. oral body temperature, between 35.0°C and 37.5°C
2. systolic blood pressure, 90 to 140 mm Hg
3. diastolic blood pressure, 45 to 90 mm Hg
4. pulse rate, 40 to 100 bpm

   * Female subjects must be:

<!-- -->

1. postmenopausal (defined as 12 months with no menses, age > 40

   years and with a follicle-stimulating hormone [FSH] level of >40 u/mL, and serum E2 < 73 pmol/L), or
2. surgically sterilized at least 3 months prior to baseline (eg, documented

   hysterectomy or tubal ligation), or
3. premenopausal and if unsterilized must have used a medically

   accepted method of contraception for 3 months (or abstained from

   sexual intercourse) prior to the screening period, and agree to use a

   medically accepted method of contraception during the trial (including

   the screening period prior to receiving trial medication) and for

   2 months after stopping the trial medication. An acceptable method of

   contraception includes one of the following:

i. stable oral, transdermal, injectable, or sustained-release vaginal

hormonal contraceptive regimen without breakthrough uterine

bleeding for 3 months prior to Screening; in addition, during

study use of condom and/or spermicide (when marketed in the

country).

ii. intrauterine device (inserted at least 2 months prior to Screening

visit); in addition, during study use of condom and/or spermicide

(when marketed in the country).

iii. condom (male or female) with spermicide (when marketed

within the country),

iv. diaphragm or cervical cap with spermicide (when marketed

within the country) and condom (male),

- Non-vasectomized men must agree to use a condom with spermicide or abstain from sexual intercourse, during the trial and for 1 month after stopping the medication.

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant (within

  3 months of ending the study), or are breastfeeding.
* Subjects who, in the opinion of the investigator, will not be able to participate optimally in the study.
* Any surgical or medical condition which might significantly alter the

absorption, distribution, metabolism or excretion of any drug. The investigator

should be guided by evidence of any of the following, and be discussed with

the sponsor prior to enrollment into the trial:

1. history or presence of inflammatory bowel disease, ulcers,

   gastrointestinal or rectal bleeding;
2. history of major gastrointestinal tract surgery such as gastrectomy,

   gastroenterostomy, or bowel resection;
3. history of pancreatic injury or pancreatitis;
4. history or presence of liver disease or liver injury;
5. history or presence of impaired renal function as indicated by clinically

   significant elevation in creatinine, blood urea nitrogen [BUN]/urea, urinary albumin, or

   clinically significant urinary cellular constituents ; or
6. history of urinary obstruction or difficulty in voiding.

   - Subject who has a history of any infectious disease within 4 weeks prior to

   drug administration that in the opinion of the investigator, affects the subject's ability to participate in the trial.
   * Subjects who are positive for hepatitis B surface antigen, hepatitis C

   antibodies or human immunodeficiency virus [HIV].

   - Subjects who have a positive screen for drugs with a high potential for abuse

   (during the Screening period or clinical conduct of the trial).

   - Subjects with a history of psychiatric or personality disorders that in the

   opinion of the investigator and sponsor, affects the subject's ability to

   participate in the trial.

   - Subjects with a history of alcohol or drug abuse in the past 2 years.- Subjects who have donated blood in the past 60 days.

   - Subjects who have previously received boceprevir.
   * Subjects who are currently participating in another clinical study or have

   participated in a clinical study (e.g., laboratory or clinical evaluation) within 30 days of baseline.

   - Subjects who are part of the study staff personnel or family members of the

   study staff personnel.
   * Subjects who have demonstrated allergic reactions (eg, food, drug, atopic

   reactions or asthmatic episodes) which, in the opinion of the investigator and

   sponsor, interfere with their ability to participate in the trial.

   - Subjects who smoke more than 10 cigarettes or equivalent tobacco use per

   day.
   * Subjects who have a history of malignancy.
   * Subjects who have received any prohibited treatment (prescription and non prescription medication except acetaminophen, potent inhibitors and inducers of cytochrome P3A [CYP3A4], or vitamins and herbals) more recently than the indicated washout period prior to Randomization which, in the opinion of the investigator and sponsor, interferes with their ability to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Boceprevir Tablets Then Capsules ( Fed): Participants will start therapy with a single dose of boceprevir tablets, orally, in fed condition, and then 4 days later will take a single dose of boceprevir capsules, orally, in fed condition.
- Boceprevir Capsules Then Tablets ( Fed): Participants will start therapy with a single dose of boceprevir capsules, orally, in fed condition, and then 4 days later will take a single dose of boceprevir tablets, orally, in fed condition.
- Boceprevir Tablets Then Capsules (Fasted): Participants will start therapy with a single dose of boceprevir tablets, orally, following an overnight fast and then 4 days later will receive a single dose of boceprevir capsules, orally, following and overnight fast.
- Boceprevir Capsules Then Tablets (Fasted): Participants will start therapy with a single dose of boceprevir capsules, orally, following an overnight fast and then 4 days later will receive a single dose of boceprevir tablets, orally, following and overnight fast.
Period: Period 1, Fed (Part 1)
Arm/Group | Boceprevir Tablets Then Capsules ( Fed) | Boceprevir Capsules Then Tablets ( Fed) | Boceprevir Tablets Then Capsules (Fasted) | Boceprevir Capsules Then Tablets (Fasted)
Started | 30 | 30 | 0 | 0
Completed | 30 | 30 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 2, Fed (Part 1)
Arm/Group | Boceprevir Tablets Then Capsules ( Fed) | Boceprevir Capsules Then Tablets ( Fed) | Boceprevir Tablets Then Capsules (Fasted) | Boceprevir Capsules Then Tablets (Fasted)
Started | 30 | 30 | 0 | 0
Completed | 30 | 30 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 3, Fasted (Part 2)
Arm/Group | Boceprevir Tablets Then Capsules ( Fed) | Boceprevir Capsules Then Tablets ( Fed) | Boceprevir Tablets Then Capsules (Fasted) | Boceprevir Capsules Then Tablets (Fasted)
Started | 0 | 0 | 59 | 58
Completed | 0 | 0 | 59 | 58
Not Completed | 0 | 0 | 0 | 0
Period: Period 4, Fasted (Part 2)
Arm/Group | Boceprevir Tablets Then Capsules ( Fed) | Boceprevir Capsules Then Tablets ( Fed) | Boceprevir Tablets Then Capsules (Fasted) | Boceprevir Capsules Then Tablets (Fasted)
Started | 0 | 0 | 59 | 58
Completed | 0 | 0 | 58 | 58
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boceprevir Tablets Then Capsules (Fed) | Boceprevir Capsules Then Tablets (Fed) | Boceprevir Tablets Then Capsules (Fasted) | Boceprevir Capsules Then Tablets (Fasted) | Total
Number analyzed (Participants) | 30 | 30 | 59 | 58 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 59 | 58 | 177
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 27 | 39 | 94
  Male | 20 | 12 | 32 | 19 | 83

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Curve (AUC) From Hour 0 to the Final Quantifiable Sample (AUCtf) for Boceprevir Tablets Versus Capsules in Fed State
Description: AUC is the measure of total plasma exposure of a drug over a given time period. AUC is derived from the area under the plasma drug concentration-time curve.
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Groups:
- Boceprevir Tablets (Fed): In Part 1 of the study, participants received a single dose of boceprevir (800 mg) in tablet formulation in a cross-over manner during either Period 1 or Period 2 under fed conditions.
- Boceprevir Capsules (Fed): In Part 1 of the study, participants received a single dose of boceprevir (800 mg) in capsule formulation in a cross-over manner during either Period 1 or Period 2 under fed conditions.
Arm/Group | Boceprevir Tablets (Fed) | Boceprevir Capsules (Fed)
Number analyzed (Participants) | 60 | 60
ng*hr/mL | 7385 [6939 to 7859] | 6644 [6243 to 7071]
Statistical Analysis 1: Comparison: Boceprevir Tablets (Fed); Test type: Non-Inferiority or Equivalence — Comparison of boceprevir tablet versus capsule used a mixed-effects model with fixed effects for formulation, sequence, and period, and a random effect for participant within sequence. The geometric mean ratio (GMR) of boceprevir tablet to boceprevir capsule is presented with two-sided 90% CIs. Equivalence of formulations was signified by the GMR falling within prespecified bioequivalence bounds; ANOVA; Least Squares Geometric Mean Ratio = 1.11, 90% CI 2-sided [1.07 to 1.15]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Boceprevir Tablets Versus Capsules in Fed State
Description: Cmax is the highest plasma drug concentration observed on the plasma concentration-time curve.
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Arm/Group | Boceprevir Tablets (Fed) | Boceprevir Capsules (Fed)
Number analyzed (Participants) | 60 | 60
ng*hr/mL | 2161 [1993 to 2343] | 1515 [1394 to 1642]
Statistical Analysis 1: Comparison: Boceprevir Tablets (Fed) vs Boceprevir Capsules (Fed); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Least Squares Geometric mean ratio = 1.43, 90% CI 2-sided [1.32 to 1.54]

3. Primary Outcome: AUCtf for Boceprevir Tablets Versus Capsules in Fasted State
Description: as for outcome 1
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Groups:
- Boceprevir Tablets (Fasted): In Part 2 of the study, participants received a single dose of boceprevir (800 mg) in tablet formulation in a cross-over manner during either Period 3 or Period 4 under fasted conditions.
- Boceprevir Capsules (Fasted): In Part 2 of the study, participants received a single dose of boceprevir (800 mg) in capsule formulation in a cross-over manner during either Period 3 or Period 4 under fasted conditions.
Arm/Group | Boceprevir Tablets (Fasted) | Boceprevir Capsules (Fasted)
Number analyzed (Participants) | 117 | 117
ng*hr/mL | 4329 [4109 to 4561] | 3935 [3734 to 4146]
Statistical Analysis 1: Comparison: Boceprevir Tablets (Fasted) vs Boceprevir Capsules (Fasted); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Least Squares Geometric mean ratio = 1.10, 95% CI 2-sided [1.06 to 1.14]

4. Primary Outcome: Cmax of Boceprevir Tablets Versus Capsules in Fasted State
Description: Cmax is the highest plasma drug concentration observed on the plasma concentration-time curve.
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Boceprevir Tablets (Fasted) | Boceprevir Capsules (Fasted)
Number analyzed (Participants) | 117 | 117
ng/mL | 1263 [1196 to 1333] | 1103 [1044 to 1164]
Statistical Analysis 1: Comparison: Boceprevir Tablets (Fasted) vs Boceprevir Capsules (Fasted); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Least Squares Geometric mean ratio = 1.15, 90% CI 2-sided [1.09 to 1.21]

5. Primary Outcome: AUC From Hour 0 to Infinity (AUCinf) in Fed State
Description: as for outcome 1
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Arm/Group | Boceprevir Tablets (Fed) | Boceprevir Capsules (Fed)
Number analyzed (Participants) | 57 | 52
ng*hr/mL | 7457 [7014 to 7928] | 6879 [6467 to 7318]

6. Primary Outcome: AUCinf in Fasted State
Description: as for outcome 1
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Arm/Group | Boceprevir Tablets (Fasted) | Boceprevir Capsules (Fasted)
Number analyzed (Participants) | 94 | 84
ng*hr/mL | 4534 [4285 to 4798] | 4119 [3885 to 4367]

7. Primary Outcome: Half Life (t1/2) of Boceprevir in Fed State
Description: T1/2 is the time required for a given drug concentration to decrease by 50%.
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Boceprevir Tablets (Fed) | Boceprevir Capsules (Fed)
Number analyzed (Participants) | 57 | 52
hours | 1.61 (0.46) | 1.46 (0.34)

8. Primary Outcome: t1/2 Boceprevir in Fasted State
Description: T1/2 is the time required for a given drug concentration to decrease by 50%.
Time Frame: Predose through 72 hours post-dose
Population: Analysis is per protocol; all available data are included in the model. No imputation is used for missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Boceprevir Tablets (Fasted) | Boceprevir Capsules (Fasted)
Number analyzed (Participants) | 93 | 82
hours | 5.33 (0.73) | 6.39 (0.84)

ADVERSE EVENTS:
Description: In this study, participants received two single doses of boceprevir 800 mg, once as capsules and once as tablets, under fed and fasted conditions, in a crossover manner; adverse events were pooled as tablets (fed condition), capsules (fed condition), tablets (fasted condition), or capsules (fasted condition).
Arm/Group | Boceprevir Tablets (Fed) | Boceprevir Capsules (Fed) | Boceprevir Tablets (Fasted) | Boceprevir Capsules (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/117 | 0/117
Other Adverse Events (participants affected / at risk) | 13/60 | 6/60 | 7/117 | 5/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir Tablets (Fed) (N=60) | Boceprevir Capsules (Fed) (N=60) | Boceprevir Tablets (Fasted) (N=117) | Boceprevir Capsules (Fasted) (N=117)
Abdominal pain lower (Gastrointestinal disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 4 (4) | 7 (7) | 5 (5)
Menstruation irregular (Reproductive system and breast disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication. The sponsor shall have the right to review and comment.